CLINICAL TRIAL: NCT04611074
Title: Health-related Quality of Life and Symptom Burden in Patients at Nordic Clinic Before, During and After Personalised, Functional Medicine Treatments and Lifestyle Interventions
Brief Title: Health-related Quality of Life in Patients at Nordic Clinic
Status: Terminated | Type: Observational
Why Stopped: Technical and recruitment issues.
Sponsor: Nordic Clinic Stockholm (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Sponsor
Other Study IDs: HRQL1
Record Dates: First submitted 2019-08-30; First posted 2020-11-02 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Chronic Disease
Keywords: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nordic Clinic is a private clinic for personalised treatment based on the Functional Medicine concept. In summary, functional medicine is aimed at addressing the lifestyle and behavioral factors that are believed to contribute to the symptoms the patient suffers from. In short, the treatment is based on a timeline of health-related life events, current lifestyle factors and behaviors and physiological examinations to develop a personalised lifestyle program. The main component of the treatment provided at Nordic Clinic is in-depth lifestyle coaching to achieve the desired behavioral and lifestyle changes.

Working at the clinic is a clinical physiologist, nutritionist, physician specialist in general medicine and researchers work. The vast majority of people who apply for the clinic have long-standing symptoms that have been investigated by the healthcare system without any organic explanation for the symptoms having been identified. Common causes are gastrointestinal problems, persistent fatigue and insomnia. The aim of the study is to investigate symptom-borne and health-related quality of life during and after treatment and to identify predictors of improvement of health-related quality of life. The main purpose is to investigate whether the health-related quality of life is improved during treatment. This is an observational study and all adult patients who are able to complete the web form in Swedish at the clinic are asked to participate. Participants who give consent will receive a link to the questionnaire via email once a month for one year and once after two years. Participants are recruited for two years, and will be completed after the last questionnaire is completed by the last included participant, ie autumn 2022. In addition to the self-assessments, the number of visits to the clinic, sampling and results, who finances the treatment and treatment plan are recorded.

The first aim is to investigate improvement in symptom burden and health related quality of life during and after treatment (does symptom burden and health related quality of improve during treatment and are improvements stable at the 2 year follow-up?) The second aim is to investigate factors that predict recovery (Do persons with a high level of motivation for behavioural change experience a better improvement in symptom burden and health related quality of life than persons with a low level of motivation for behavioural change?).

DETAILED DESCRIPTION:
Research plan

Health related quality of life in patients at the Nordic Clinic

Background

Nordic Clinic is a private clinic that provides personalised treatment based on functional medicine. The vast majority of the patients seeking care at the clinic suffer from unexplained medical symptoms, most commonly fatigue and abdominal symptoms, and have previously been medically evaluated by health care. Working at the clinic are a clinical physiologist, nutritional therapist, licensed physician and a researcher. Patients follow a clinical treatment process starting with the physician progressing through to the nutritionist. Treatment is covered either by the patient themselves, by employers or health insurances.

Before treatment is initialised, an extensive medical history along with current lifestyle habits are taken. The treatment programme is based on lifestyle factors, mainly diet, sleep, stress management and physical activity. Supplements are given. Drugs are prescribed sparsely and by a licenced physician, and may include Rifaximin or other antibiotics for intestinal bacterial overgrowth, motility drugs for constipation, anti-parasitic drugs in case of parasite infection, and melatonin for sleep disturbances.

The components in the treatment programme have been investigated separately. Any supplements used are produced by reputable organisations and most of them have been part of the treatment routine for several years. The aims of the study is to evaluate improvement during and after treatment and to identify predictors of recovery. The goal is to understand the process of recovery with the long term goal to improve care given at the clinic.

Aim and research question

The first aim is to investigate improvement in symptom burden and health related quality of life during and after treatment (does symptom burden and health related quality of improve during treatment and are improvements stable at the 2 year follow-up?) The second aim is to investigate factors that predict recovery (Do persons with a high level of motivation for behavioural change experience a better improvement in symptom burden and health related quality of life than persons with a low level of motivation for behavioural change?).

Methods

Study population and inclusion criteria

All Swedish speaking patients (>1= 18 years) visiting the clinic will be asked to participate in the study by clinic personnel when visiting the clinic. All patients at the clinic are able to provide informed consent and to fill out online forms.

Procedure

This is an observational study where patients are followed over time in terms of symptom burden and health related quality of life. The study participants are asked to fill out forms once a month for one year counting from the first visit, and once again 2 years after baseline. Clinical data is collected from the medial record by the clinician at the end of the study.

Questionnaires

(Jylhä 2009)(K, S et al. 2003)(Westerlund, Brandt et al. 2014)(Smets, Garssen et al. 1995)(Andreasson, Wicksell et al. 2016)(Spitzer, Kroenke et al. 2006)(Spitzer, Kroenke et al. 1999)

Clinical variables

Information on diagnosis, number of visits, tests and test results, treatment programme and background information (including age, gender, lifestyle factors, readiness for change, education, occupation, social support, height and weight, blood pressure), will be collected from the medical record of the patient by the clinician at the end of the study period.

Statistics

Based on experience of these types of analyses, 150 participants would give a reasonable foundation for the statistical analyses. 300 unique patients are expected to enrol during the study inclusion period and expect 200 of these to complete at least the first year of data collection. In the main analysis of the first aim, the effect of time on questionnaire scores will be investigated using mixed effect linear regression to see to what extent symptom burden and health related quality of life is affected during treatment and to investigate the stability in any improvements. Secondly, it will be investigated it a high adherence to the treatment programme is associated with improvement. Thirdly, the level of adherence to the treatment programme will be compared between patients with predominant abdominal symptoms and patients with predominant fatigue.

In the main analysis of the second aim, readiness for change will be tested as a moderator of the effect of time on questionnaire scores. Secondly, the level of improvement will be compared between patients who self-fund the treatment programme and patients with funding from employer or health insurance.

Patients often present with a range of different symptoms. Principal component analysis will be performed in an exploratory analysis to investigate if there are subgroups within the patient population, and if these subgroups differ in terms of treatment response. Covariation over time of symptoms, health related quality of life and self-rated health will be investigated in exploratory analyses.

Ethical considerations

The present study poses little risk to the participant. The treatment programme that the participant would undergo independently of the study is considered safe with few and mild side effects such as rash. As part of the study the participant report health information on a web questionnaire. Health data is sensitive information and the same platform will be used as for all other data collected by the clinic for treatment. The platform that is used is certified safe (add information) and complies to the GDPR regulation.

Risk of missing serious diagnoses

When dealing with symptoms such as persistent fatigue there is a risk that serious conditions such as cancer might be missed. However, the risk is estimated as low as low as in primary care at a Vårdcentral. Our medical doctor is still active in primary health care in parallel to Nordic Clinic and has many years of experience. Most of the patients at Nordic Clinic have been thoroughly investigated in the primary care system before signing up as patients at Nordic Clinic. Should patients however present with symptoms that warrant the investigation of serious conditions like malignancies, it is made sure that a thorough investigation has indeed been performed. If it has not, our medical doctor refers them back to primary or specialist health care.

Importance

There has not been a strong research tradition to evaluate treatment programmes based on functional medicine, albeit the individual components therein have all been evaluated and are found to be safe. However, all treatments given to patients need continuing evaluation. This two-year observational study will provide information regarding treatment outcomes and stability thereof over time, in addition to identifying patient groups that get the most benefit of the treatment. Future randomised controlled trials are needed to evaluate the effectiveness of the treatment programme.

ELIGIBILITY:
Inclusion Criteria:

* All Swedish speaking patients (>/= 18 years) visiting the clinic will be asked to participate in the study by clinic personnel when they are visiting the clinic. All patients at the clinic are able to provide informed consent and to fill out online forms.

Exclusion Criteria:

* <18 years, non-Swedish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Swedish speaking patients (>1= 18 years) visiting the clinic will be asked to participate in the study by clinic personnel when they are visiting the clinic. All patients at the clinic are able to provide informed consent and to fill out online forms.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal discomfort from baseline as assessed by the Gastrointestinal Symptom Rating Scale for IBS questionnaire (GSRS-IBS) | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  Self-reported satiety, abdominal pain, diarrhoea, constipation and bloating is measured with GSRS-IBS with the following outcomes: No discomfort at all, Minor discomfort, Mild discomfort, Moderate discomfort, Moderately severe discomfort, Severe discomfort, Very severe discomfort.
Change in fatigue from baseline as assessed by the Multidimensional Fatigue Inventory | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  General fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue is evaluated on a scale from 1-5, where 1 is true and 5 is not true.
Change in health-related quality of life from baseline as assessed by the 36-Item Short Form Health Survey (SF-36) | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  The SF-36 measures physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.
Change in sleep from baseline as assessed by the Karolinska Sleep Questionnaire (KSQ) | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  KSQ is a self-assessment form that measures difficulty falling asleep, disturbed sleep, repeated awakenings, early wakings, difficulty waking up, insufficient rest during the night, nightmares, snoring, daytime effects. The questionnaire contains 13 questions about sleep and sleepiness which are answered according to a five-point scale from 1 (never/very good) to 5 (always/very bad).
Change in anxiety from baseline as assessed by the Generalised Anxiety Disorder 7-item scale (GAD-7) | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  GAD-7 is a self-assessment form that measures seven anxiety-related symptoms using the following scale: Not at all (0), Several days (1), More than half the days (2), Nearly every day (3).
Change in presence or severity of depression from baseline as assessed by the Patient Health Questionnaire-9 (PHQ-9) | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  PHQ-9 screens for presence or severity of depression according to the DSM-IV criteria. It measures nine depression-related symptoms using the following scale: Not at all (0), Several days (1), More than half the days (2), Nearly every day (3).
Change in overall health from baseline as assessed by the Self-rated health questionnaire | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  The self-rated health questionnaire is a single question questionnaire, evaluating overall health at the time of the survey using the scale very good" (1), "good" (2), "moderate" (3), "bad" (4) or "very bad" (5).

SECONDARY OUTCOMES:
Correlation between motivation for behavioral change and change in symptom burden and health-related quality of life | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  Correlation between motivation for behavioral change and change in the primary outcome measures
Predictability of the predominance of fatigue or abdominal-related symptomatology for adherence to the treatment programme | Baseline (time of enrollment), then each month 1-12 months after baseline, and then at 24 months.
  Correlation between outcome measures in Gastrointestinal Symptom Rating Scale for IBS questionnaire (GSRS-IBS) and adherence to the treatment programme.

CONTACTS AND LOCATIONS:
Overall Officials: Annie ML Pettersson, PhD, Principal Investigator — Nordic Clinic
Locations (1):
- Nordic Clinic, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andreasson A, Wicksell RK, Lodin K, Karshikoff B, Axelsson J, Lekander M. A global measure of sickness behaviour: Development of the Sickness Questionnaire. J Health Psychol. 2018 Sep;23(11):1452-1463. doi: 10.1177/1359105316659917. Epub 2016 Jul 24. PMID 27458105
- [Background] Bryant PA, Trinder J, Curtis N. Sick and tired: Does sleep have a vital role in the immune system? Nat Rev Immunol. 2004 Jun;4(6):457-67. doi: 10.1038/nri1369. No abstract available. PMID 15173834
- [Background] Hallgren M, Stubbs B, Vancampfort D, Lundin A, Jaakallio P, Forsell Y. Treatment guidelines for depression: Greater emphasis on physical activity is needed. Eur Psychiatry. 2017 Feb;40:1-3. doi: 10.1016/j.eurpsy.2016.08.011. Epub 2016 Nov 10. No abstract available. PMID 27837666
- [Background] Jylha M. What is self-rated health and why does it predict mortality? Towards a unified conceptual model. Soc Sci Med. 2009 Aug;69(3):307-16. doi: 10.1016/j.socscimed.2009.05.013. Epub 2009 Jun 10. PMID 19520474
- [Background] Wiklund IK, Fullerton S, Hawkey CJ, Jones RH, Longstreth GF, Mayer EA, Peacock RA, Wilson IK, Naesdal J. An irritable bowel syndrome-specific symptom questionnaire: development and validation. Scand J Gastroenterol. 2003 Sep;38(9):947-54. doi: 10.1080/00365520310004209. PMID 14531531
- [Background] Rezaie A, Pimentel M, Rao SS. How to Test and Treat Small Intestinal Bacterial Overgrowth: an Evidence-Based Approach. Curr Gastroenterol Rep. 2016 Feb;18(2):8. doi: 10.1007/s11894-015-0482-9. PMID 26780631
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Westerlund A, Brandt L, Harlid R, Akerstedt T, Lagerros YT. Using the Karolinska Sleep Questionnaire to identify obstructive sleep apnea syndrome in a sleep clinic population. Clin Respir J. 2014 Oct;8(4):444-54. doi: 10.1111/crj.12095. PMID 25396257
- [Background] Younge JO, Gotink RA, Baena CP, Roos-Hesselink JW, Hunink MG. Mind-body practices for patients with cardiac disease: a systematic review and meta-analysis. Eur J Prev Cardiol. 2015 Nov;22(11):1385-98. doi: 10.1177/2047487314549927. Epub 2014 Sep 16. PMID 25227551